CLINICAL TRIAL: NCT02271594
Title: Treating Diabetic Lipohypertrophy With Intensive Education Versus Standard Care: A Randomized, Prospective, Controlled Study in Ealing, United Kingdom
Brief Title: Treating Diabetic Lipohypertrophy With Intensive Education Versus Standard Care
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Becton, Dickinson and Company (Industry)
Collaborators: Ealing Hospital NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DBC-14LIPOINJ02
Record Dates: First submitted 2014-10-20; First posted 2014-10-22 (Estimated); Results first posted 2021-06-09 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-06

CONDITIONS: Insulin Injections and Lipohypertrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Active Comparator): Intensive education on injection technique
  Interventions: Behavioral: Intensive Training on Best Insulin Injection Technique
- Control (Placebo Comparator): Standard education on injection technique
  Interventions: Behavioral: Standard education on injection technique

INTERVENTIONS:
Behavioral: Intensive Training on Best Insulin Injection Technique — The intervention consists of instructing patients in whom LH is detected and who are currently injecting into it to move injections to non-LH areas; reducing insulin doses initially by 10-20% to avoid hypoglycaemia and then titrating to target control; instructing these patients to correctly rotate sites (leaving 1 cm between injection punctures and allowing used sites to heal for 2-4 weeks before injecting in them again); instructing these patients to forego needle reuse; and instructing these patients to switch to 4 mmx32G needles. A battery of tools (described below) will be used to deliver and reinforce this training, including frequent contact by phone or other electronic means after the initial training.
  Other Names: Standard education on injection technique
  Arms: Intervention
Behavioral: Standard education on injection technique — Usual and customary education and training normally provided injecting patients at the center
  Arms: Control

SUMMARY:
The investigators intend to assess the impact of optimized injection technique on the evolution of clinical parameters in insulin-treated patients with diabetes (DM) who have clinical lipohypertrophy (LH) in a controlled, prospective study with a follow-up of 6 months, conducted at Ealing Hospital, West London, UK. DM patients who have LH and inject into it will be randomized to either switch to normal tissue sites with intensive education as to why and how and use of a 4mm pen needle, or to continue with standard care. The endpoints measured will include the impact on glucose control parameters, consumption of insulin, hypoglycaemia rates, use of health services resources and health care costs

DETAILED DESCRIPTION:
This is an interventional clinical trial at Ealing Hospital (UK) in patients with DM1 and DM2 treated with insulin for at least 1 year, aged from 18 to 75 years inclusive, with a goal of 95 patients randomized to the 'LH+ Intervention' arm and 95 patients randomized to the 'LH+ Standard Care' arm. LH+ refers to the presence of clinically-confirmed LH about which there is little or no doubt as to its presence. The study takes place over 4 clinic visits, which form part of their usual clinical visits (spaced at 3-month intervals in Ealing). Each visit is described below.

INTERVENTION The intervention consists of instructing patients in whom LH is detected and who are currently injecting into it to move injections to non-LH areas; reducing insulin doses initially by 10-20% to avoid hypoglycaemia and then titrating to target control; instructing these patients to correctly rotate sites (leaving 1 cm between injection punctures and allowing used sites to heal for 2-4 weeks before injecting in them again); instructing these patients to forego needle reuse; and instructing these patients to switch to 4 mmx32G needles. A battery of tools (described below) will be used to deliver and reinforce this training, including frequent contact by phone or other electronic means after the initial training.

CONTROL Standard care means affording the patients randomized to the control arm the customary education and follow-up usually given at the centre. This would include appraising them of the presence of LH (if they were not previously aware) and stating that injections should not be given into that area. The training approach, tools and intensive follow-up given the Intervention arm patients will not be given to the Controls. Additionally, at their return visit (3 and 6 months), Control patients will be asked if they did indeed change their injection habits (e.g. stopped injecting into LH) since entering the study. Those who did and those who did not will be analysed separately to see if there is a difference in outcomes and both groups will be compared to the Intervention arm patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with DM1 or DM2, diagnosed for more than a year from the time of inclusion
2. Age between 18 and 75 years old, inclusive
3. Treatment by insulin injection using pen injector for at least 1 year - concomitant oral therapy or GLP-1 injections are allowed
4. Self-care (patients must be giving injections to themselves as opposed to getting them by third parties)
5. Presence of LH on structured physical exam (if in doubt, the patient will not be included)
6. Injections performed frequently into the LH (at least once per day)
7. Self-monitoring of blood glucose (SMBG) and willingness to bring meter to every visit for electronic download
8. Willingness to fill out a diary recording any adverse event (e.g. hypoglycaemia, ambulance call out, unscheduled visit to health care facility) or symptoms that occur during the study
9. Ability so speak and read English or accompanied by a person who can competently translate for the patient

Exclusion Criteria:

1. Pregnancy (declarative)
2. Ongoing participation in another clinical trial
3. Conditions other than diabetes treatment which might cause lipodystrophies (ex: antiretroviral therapy)
4. Medical conditions that may, in the opinion of the PI, influence study results (ex: currently active cancer, uncontrolled endocrine disorder, eating disorders)
5. Current treatments that may, in the opinion of the PI, influence study results (ex: long-term corticosteroids)
6. Other injectable treatment in diabetes (with the exception of GLP-1) such as insulin pumps, syringes
7. Study staff will document the reasons for the exclusion, if any.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2015-01; Primary Completion 2016-08 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Grace E Vanterpool, RN, Principal Investigator — Ealing Hospital, Northwest London NHS Trust
Locations (1):
- Ealing Hospital, Middlesex, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Intensive Training: The intervention consists of instructing patients in whom lipohypertrophy (LH) is detected and who are currently injecting into it to move injections to non-LH areas; reducing insulin doses initially by 10-20% to avoid hypoglycaemia and then titrating to target control; instructing these patients to correctly rotate sites (leaving 1 cm between injection punctures and allowing used sites to heal for 2-4 weeks before injecting in them again); instructing these patients to forego needle reuse; and instructing these patients to switch to 4 mmx32G needles. A battery of tools (described below) will be used to deliver and reinforce this training, including frequent contact by phone or other electronic means after the initial training.
- Standard Care: Standard care means affording the patients randomized to the control arm the customary education and follow-up usually given at the centre. This would include appraising them of the presence of LH (if they were not previously aware) and stating that injections should not be given into that area. The training approach, tools and intensive follow-up given the Intervention arm patients will not be given to the Controls. Additionally, at their return visit (3 and 6 months), Control patients will be asked if they did indeed change their injection habits (e.g. stopped injecting into LH) since entering the study. Those who did and those who did not will be analysed separately to see if there is a difference in outcomes and both groups will be compared to the Intervention arm patients.
Period: Overall Study
Arm/Group | Intensive Training | Standard Care
Started | 19 | 12
Completed | 0 (Study closed down) | 0 (Study closed down)
Not Completed | 19 | 12
Not completed — Study closed; recruiting failure | 19 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intensive Training | Standard Care | Total
Number analyzed (Participants) | 19 | 12 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (12) | 53 (13) | 52 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 12 | 5 | 17

OUTCOME MEASURES:

1. Primary Outcome: HbA1c
Description: The mean HbA1c from baseline to be compared to six months
Time Frame: 6 months
Population: Study terminated prior to study endpoint; no 6-month data were collected
Arm/Group | Intensive Training | Standard Care
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Blood Glucose (BG) Values
Description: Number of BG values within target range
Time Frame: 6 months
Population: Data were not collected
Arm/Group | Intervention | Control
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Hypoglycemia Reactions
Description: Number and severity of hypoglycemic reactions
Time Frame: 6 months
Population: Not recorded
Arm/Group | Intensive Training | Standard Care
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Total Daily Dose (TDD) of Insulin
Description: The mean TDD from baseline to be compared to six months
Time Frame: 6 months
Population: Not recorded
Arm/Group | Intensive Training | Standard Care
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Health Care Costs
Description: The mean health care costs from baseline to be compared to six months
Time Frame: 6 months
Population: Not recorded
Arm/Group | Intensive Training | Standard Care
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 18 months
Groups:
- Intensive Training: The intervention consists of instructing patients in whom lipohypertrophy (LH) is detected and who are currently injecting into it to move injections to non-LH areas; reducing insulin doses initially by 10-20% to avoid hypoglycaemia and then titrating to target control; instructing these patients to correctly rotate sites (leaving 1 cm between injection punctures and allowing used sites to heal for 2-4 weeks before injecting in them again); instructing these patients to forego needle reuse; and instructing these patients to switch to 4 mmx32G needles. A battery of tools (described below) will be used to deliver and reinforce this training, including frequent contact by phone or other electronic means after the initial training.
  Intensive Training on Best Insulin Injection Technique: The intervention consists of instructing patients in whom LH is detected and who are currently injecting into it to move injections to non-LH areas; reducing insulin doses initially by 10-20%
Arm/Group | Intensive Training | Standard Care
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/12
Other Adverse Events (participants affected / at risk) | 0/19 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No